CLINICAL TRIAL: NCT05444556
Title: The Effect of Imlunestrant on CYP2C8, CYP2C19, CYP2D6, P-gp, and BCRP Activity and the Effect of P-gp Inhibition on Imlunestrant Pharmacokinetics in Healthy Women of Non-childbearing Potential
Brief Title: A Study of Imlunestrant (LY3484356) in Female Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18413; J2J-MC-JZLI (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11-15

CONDITIONS: Healthy
MeSH Terms: interventions — Imlunestrant; repaglinide; Omeprazole; Dextromethorphan; Quinidine; Rosuvastatin Calcium; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Imlunestrant + Repaglinide (Cohort 1) (Experimental): Participants received:
  Day 1: A single oral dose of 0.5 mg repaglinide administered alone. Day 3: A single oral dose of 800 mg imlunestrant, followed approximately 2 hours later by 0.5 mg repaglinide, both administered orally.
  Interventions: Drug: Imlunestrant; Drug: Repaglinide
- mlunestrant + Omeprazole & Dextromethorphan (Cohort 2) (Experimental): Participants received:
  Day 1: A single oral dose of 20 mg omeprazole and 30 mg dextromethorphan, administered in the morning.
  Day 3: A single oral dose of 800 mg imlunestrant, followed immediately by 20 mg omeprazole and 30 mg dextromethorphan, all administered orally.
  Interventions: Drug: Imlunestrant; Drug: Omeprazole; Drug: Dextromethorphan
- Imlunestrant + Quinidine (Cohort 3) (Experimental): Participants received:
  Day 1: A single oral dose of 400 mg imlunestrant, administered in the morning. Days 15 to 17 and 19 to 24: Twice-daily oral doses of 200 mg quinidine, administered alone.
  Day 18: A single oral dose of 400 mg imlunestrant administered in combination with 200 mg quinidine (quinidine was dosed twice on this day as part of the regular regimen).
  Interventions: Drug: Imlunestrant; Drug: Quinidine
- Imlunestrant + Rosuvastatin & Digoxin (Cohort 4) (Experimental): Participants received:
  Day 1: A single oral dose of 10 mg rosuvastatin and 0.25 mg digoxin, administered in the morning.
  Day 10: A single oral dose of 400 mg imlunestrant, administered in combination with 10 mg rosuvastatin and 0.25 mg digoxin, all administered orally.
  Interventions: Drug: Imlunestrant; Drug: Rosuvastatin; Drug: Digoxin

INTERVENTIONS:
Drug: Imlunestrant — Administered orally.
  Other Names: LY3484356
Drug: Repaglinide — Administered orally.
  Arms: Imlunestrant + Repaglinide (Cohort 1)
Drug: Omeprazole — Administered orally.
  Arms: mlunestrant + Omeprazole & Dextromethorphan (Cohort 2)
Drug: Dextromethorphan — Administered orally.
  Arms: mlunestrant + Omeprazole & Dextromethorphan (Cohort 2)
Drug: Quinidine — Administered orally.
  Arms: Imlunestrant + Quinidine (Cohort 3)
Drug: Rosuvastatin — Administered orally.
  Arms: Imlunestrant + Rosuvastatin & Digoxin (Cohort 4)
Drug: Digoxin — Administered orally.
  Arms: Imlunestrant + Rosuvastatin & Digoxin (Cohort 4)

SUMMARY:
The main purpose of this study is to evaluate the effect of imlunestrant on repaglinide, omeprazole and dextromethorphan, and rosuvastatin and digoxin. The study will also investigate the effect of quinidine on imlunestrant in female healthy participants of non-childbearing potential. The safety and tolerability of imlunestrant will be investigated in female healthy participants of non-childbearing potential. The study will last approximately up to 32 days for each participant excluding the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical assessment
* Body mass index (BMI) within the range 18.0 to 35.0 kilograms per meter squared (kg/m²)
* Female participants of non childbearing potential.

Exclusion Criteria:

* Have known allergies to imlunestrant, related compounds or any components of the formulation, repaglinide, omeprazole, dextromethorphan, quinidine, rosuvastatin, or digoxin, as appropriate, or history of significant atopy.
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing
* Use or intend to use any prescription medications/products within 14 days prior to first dose until completion of the follow-up visit, unless deemed acceptable by the investigator (or designee), including but not limited to medications that inhibit or induce cytochrome P450 (CYP) 2C8, CYP2C19, CYP2D6, P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 113 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Altasciences Clinical Los Angeles, Inc, Cypress, California
  - Qps-Mra, Llc, South Miami, Florida
  - ICON Early Phase Services, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Imlunestrant + Omeprazole & Dextromethorphan (Cohort 2): Participants received:
  Day 1: A single oral dose of 20 mg omeprazole and 30 mg dextromethorphan, administered in the morning.
  Day 3: A single oral dose of 800 mg imlunestrant, followed immediately by 20 mg omeprazole and 30 mg dextromethorphan, all administered orally.
Period: Overall Study
Arm/Group | Imlunestrant + Repaglinide (Cohort 1) | Imlunestrant + Omeprazole & Dextromethorphan (Cohort 2) | Imlunestrant + Quinidine (Cohort 3) | Imlunestrant + Rosuvastatin & Digoxin (Cohort 4)
Started | 27 | 27 | 32 | 27
Received at Least One Dose of Study Drug | 27 | 27 | 32 (One participant did not receive the second dose of imlunestrant in combination with quinidine on Day 18, or the subsequent doses of quinidine alone on Days 19 through 24) | 27 (One participant did not receive the planned dose of imlunestrant in combination with rosuvastatin and digoxin on Day 10.)
Completed | 27 | 27 | 30 | 26
Not Completed | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Imlunestrant + Repaglinide (Cohort 1) | Imlunestrant + Omeprazole & Dextromethorphan (Cohort 2) | Imlunestrant + Quinidine (Cohort 3) | Imlunestrant + Rosuvastatin & Digoxin (Cohort 4) | Total
Number analyzed (Participants) | 27 | 27 | 32 | 27 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (8.2) | 52.6 (8.2) | 55.9 (6.3) | 54.1 (7.1) | 54.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 32 | 27 | 113
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 19 | 23 | 14 | 78
  Not Hispanic or Latino | 5 | 8 | 9 | 13 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 4 | 7 | 19
  White | 23 | 21 | 27 | 19 | 90
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 27 | 32 | 27 | 113

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Repaglinide (Cohort 1)
Description: PK: AUC[0-∞] of Repaglinide
Time Frame: Day 1 and Day 3: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Population: All participants in Cohort 1 who received at least one dose of repaglinide and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- 0.5 mg Repaglinide: Participants received a single oral dose of 0.5 mg repaglinide administered alone on Day 1.
- 800 mg Imlunestrant + 0.5 mg Repaglinide: Participants received a single oral dose of 800 mg imlunestrant, followed approximately 2 hours later by 0.5 mg repaglinide, both administered orally on Day 3.
Arm/Group | 0.5 mg Repaglinide | 800 mg Imlunestrant + 0.5 mg Repaglinide
Number analyzed (Participants) | 24 | 23
nanogram*hour per milliliter (ng*hr/mL) | 13.0 (31) | 13.6 (31)

2. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Repaglinide (Cohort 1)
Description: PK: Cmax of Repaglinide
Time Frame: Day 1 and Day 3: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Population: All participants in Cohort 1 who received at least one dose of repaglinide and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | 0.5 mg Repaglinide | 800 mg Imlunestrant + 0.5 mg Repaglinide
Number analyzed (Participants) | 27 | 27
nanogram per millilitre (ng/mL) | 10.5 (38) | 9.84 (44)

3. Primary Outcome: PK: AUC[0-∞] of Omeprazole (Cohort 2)
Description: PK: AUC[0-∞] of Omeprazole
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8,12, and 24 h postdose; Day 3: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, and 48 h postdose
Population: All participants in Cohort 2, who received at least one dose of omeprazole and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 20 mg Omeprazole + 30 mg Dextromethorphan: Participants received a single oral dose of 20 mg omeprazole and 30 mg dextromethorphan, administered in the morning on Day 1
- 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan: Participants received a single oral dose of 800 mg imlunestrant, followed immediately by 20 mg omeprazole and 30 mg dextromethorphan, all administered orally on Day 3.
Arm/Group | 20 mg Omeprazole + 30 mg Dextromethorphan | 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan
Number analyzed (Participants) | 21 | 26
ng*hr/mL | 703 (77) | 825 (74)

4. Primary Outcome: PK: Cmax of Omeprazole (Cohort 2)
Description: PK: Cmax of Omeprazole
Time Frame: as for outcome 3
Population: All participants in Cohort 2, who received at least one dose of omeprazole and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 20 mg Omeprazole + 30 mg Dextromethorphan | 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan
Number analyzed (Participants) | 27 | 27
ng/mL | 316 (73) | 405 (57)

5. Primary Outcome: PK: AUC[0-∞] of Omeprazole Metabolite: 5-hydroxyomeprazole (Cohort 2)
Description: 5-hydroxyomeprazole is a major metabolite of omeprazole.
Time Frame: as for outcome 3
Population: All participants in Cohort 2, who received at least one dose of omeprazole and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 20 mg Omeprazole + 30 mg Dextromethorphan | 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan
Number analyzed (Participants) | 24 | 26
ng*hr/mL | 571 (26) | 592 (19)

6. Primary Outcome: PK: Cmax of Omeprazole Metabolite: 5-hydroxyomeprazole (Cohort 2)
Description: 5-hydroxyomeprazole is a major metabolite of omeprazole.
Time Frame: as for outcome 3
Population: All participants in Cohort 2, who received at least one dose of omeprazole and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 20 mg Omeprazole + 30 mg Dextromethorphan | 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan
Number analyzed (Participants) | 27 | 27
ng/mL | 200 (52) | 230 (42)

7. Primary Outcome: PK: AUC[0-∞] of Dextromethorphan (Cohort 2)
Description: PK: AUC[0-∞] of Dextromethorphan
Time Frame: as for outcome 3
Population: All Cohort 2 participants who received at least one dose of dextromethorphan and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 20 mg Omeprazole + 30 mg Dextromethorphan | 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan
Number analyzed (Participants) | 25 | 12
ng*hr/mL | 14.7 (127) | 16.1 (111)

8. Primary Outcome: PK: Cmax of Dextromethorphan (Cohort 2)
Description: PK: Cmax of Dextromethorphan
Time Frame: as for outcome 3
Population: All Cohort 2 participants who received at least one dose of dextromethorphan and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 20 mg Omeprazole + 30 mg Dextromethorphan | 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan
Number analyzed (Participants) | 26 | 12
ng/mL | 0.864 (124) | 1.13 (124)

9. Primary Outcome: PK: Area Under the Concentration Versus Time Curve (AUC) From Time Zero to Tlast (AUC[0-tlast]) of Dextromethorphan Metabolite: Dextrorphan (Cohort 2)
Description: Dextrorphan is a major metabolite of Dextromethorphan.
Time Frame: as for outcome 3
Population: All Cohort 2 participants who received at least one dose of dextromethorphan and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 20 mg Omeprazole + 30 mg Dextromethorphan | 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan
Number analyzed (Participants) | 26 | 26
ng*hr/mL | 11.8 (62) | 11.9 (75)

10. Primary Outcome: PK: Cmax of Dextromethorphan Metabolite: Dextrorphan (Cohort 2)
Description: Dextrorphan is a major metabolite of Dextromethorphan.
Time Frame: as for outcome 3
Population: All Cohort 2 participants who received at least one dose of dextromethorphan and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 20 mg Omeprazole + 30 mg Dextromethorphan | 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan
Number analyzed (Participants) | 26 | 26
ng/mL | 1.79 (50) | 1.97 (56)

11. Primary Outcome: PK: AUC[0-∞] of Imlunestrant (Cohort 3)
Description: PK: AUC[0-∞] of Imlunestrant
Time Frame: Day 1 and Day 18: Predose, 1, 2, 3, 4, 5, 6 ,8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 h post dose
Population: All cohort 3 participants who received at least one dose of imlunestrant and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 400 mg Imlunestrant (Day 1): Participants received a single oral dose of 400 mg imlunestrant administered alone on Day 1.
- 400 mg Imlunestrant + 200 mg Quinidine BID (Day 18): Participants received a single oral dose of 400 mg imlunestrant administered in combination with 200 mg quinidine (quinidine was dosed twice on this day as part of the regular regimen) on day 18.
Arm/Group | 400 mg Imlunestrant (Day 1) | 400 mg Imlunestrant + 200 mg Quinidine BID (Day 18)
Number analyzed (Participants) | 30 | 31
ng*hr/mL | 1970 (66) | 1870 (87)

12. Primary Outcome: PK: Cmax of Imlunestrant (Cohort 3)
Description: PK: Cmax of Imlunestrant
Time Frame: Day 1 and Day 18: Predose, 1, 2, 3, 4, 5, 6 ,8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 h post dose
Population: All cohort 3 participants who received at least one dose of imlunestrant and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 400 mg Imlunestrant (Day 1) | 400 mg Imlunestrant + 200 mg Quinidine BID (Day 18)
Number analyzed (Participants) | 32 | 31
ng/mL | 61.0 (82) | 54.3 (81)

13. Primary Outcome: PK: AUC[0-∞] of Rosuvastatin (Cohort 4)
Description: PK: AUC[0-∞] of Rosuvastatin
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, and 96 h post dose; Day 10: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, and 120 h post dose
Population: All cohort 4 participants who received at least one dose of rosuvastatin and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 10 mg Rosuvastatin + 0.25 mg Digoxin: Participants received a single oral dose of 10 mg rosuvastatin and 0.25 mg digoxin on Day 1.
- 400 mg Imlunestrant + 10 mg Rosuvastatin + 0.25 mg Digoxin: Participants received a single oral dose of 400 mg imlunestrant, administered in combination with 10 mg rosuvastatin and 0.25 mg digoxin, all administered orally on Day 10.
Arm/Group | 10 mg Rosuvastatin + 0.25 mg Digoxin | 400 mg Imlunestrant + 10 mg Rosuvastatin + 0.25 mg Digoxin
Number analyzed (Participants) | 14 | 20
ng*hr/mL | 29.0 (47) | 44.9 (51)

14. Primary Outcome: PK: Cmax of Rosuvastatin (Cohort 4)
Description: PK: Cmax of Rosuvastatin
Time Frame: as for outcome 13
Population: All cohort 4 participants who received at least one dose of rosuvastatin and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 10 mg Rosuvastatin + 0.25 mg Digoxin | 400 mg Imlunestrant + 10 mg Rosuvastatin + 0.25 mg Digoxin
Number analyzed (Participants) | 26 | 25
ng/mL | 2.99 (53) | 5.08 (59)

15. Primary Outcome: PK: AUC[0-∞] of Digoxin (Cohort 4)
Description: PK: AUC[0-∞] of Digoxin
Time Frame: as for outcome 13
Population: All cohort 4 participants who received at least one dose of digoxin and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 10 mg Rosuvastatin + 0.25 mg Digoxin | 400 mg Imlunestrant + 10 mg Rosuvastatin + 0.25 mg Digoxin
Number analyzed (Participants) | 11 | 18
ng*hr/mL | 20.2 (23) | 28.0 (19)

16. Primary Outcome: PK: Cmax of Digoxin (Cohort 4)
Description: PK: Cmax of Digoxin
Time Frame: as for outcome 13
Population: All cohort 4 participants who received at least one dose of digoxin and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 10 mg Rosuvastatin + 0.25 mg Digoxin | 400 mg Imlunestrant + 10 mg Rosuvastatin + 0.25 mg Digoxin
Number analyzed (Participants) | 25 | 25
ng/mL | 1.17 (39) | 1.88 (38)

ADVERSE EVENTS:
Time Frame: Cohort 1: up to 11 days, Cohort 2: up to 12 days, Cohort 3: up to 32 days, Cohort 4: up to 22 days
Description: All participants who received at least one dose of study drug and have at least one post dose safety assessment. Based on the planned safety analysis, adverse events were collected per dose level of treatment regimen
Groups:
- 0.5 mg Repaglinide: Cohort 1: Participants received a single oral dose of 0.5 mg repaglinide administered alone on Day 1.
- 800 mg Imlunestrant + 0.5 mg Repaglinide: Cohort 1: Participants received a single oral dose of 800 mg imlunestrant, followed approximately 2 hours later by 0.5 mg repaglinide, both administered orally on Day 3.
- 20 mg Omeprazole + 30 mg Dextromethorphan: Cohort 2: Participants received a single oral dose of 20 mg omeprazole and 30 mg dextromethorphan, administered in the morning on Day 1.
- 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan: Cohort 2: Participants received a single oral dose of 800 mg imlunestrant, followed immediately by 20 mg omeprazole and 30 mg dextromethorphan, all administered orally on Day 3.
- 400 mg Imlunestrant (Day 1): Cohort 3: Participants received a single oral dose of 400 mg imlunestrant administered alone on Day 1.
- 200 mg Quinidine BID (Days 15 to 17): Cohort 3: Participants received twice-daily oral doses of 200 mg quinidine, administered alone from days 15 to 17.
- 400 mg Imlunestrant + 200 mg Quinidine BID (Day 18): Cohort 3: Participants received a single oral dose of 400 mg imlunestrant administered in combination with 200 mg quinidine (quinidine was dosed twice on this day as part of the regular regimen) on day 18.
- 200 mg Quinidine BID (Days 19 to 24): Cohort 3: Participants received BID oral doses of 200 mg quinidine, administered alone from Days 19 to 24.
- 10 mg Rosuvastatin + 0.25 mg Digoxin: Cohort 4: Participants received a single oral dose of 10 mg rosuvastatin and 0.25 mg digoxin on Day 1.
- 400 mg Imlunestrant + 10 mg Rosuvastatin + 0.25 mg Digoxin: Cohort 4: Participants received a single oral dose of 400 mg imlunestrant, administered in combination with 10 mg rosuvastatin and 0.25 mg digoxin, all administered orally on Day 10.
Arm/Group | 0.5 mg Repaglinide: Cohort 1 | 800 mg Imlunestrant + 0.5 mg Repaglinide: Cohort 1 | 20 mg Omeprazole + 30 mg Dextromethorphan: Cohort 2 | 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan: Cohort 2 | 400 mg Imlunestrant (Day 1): Cohort 3 | 200 mg Quinidine BID (Days 15 to 17): Cohort 3 | 400 mg Imlunestrant + 200 mg Quinidine BID (Day 18): Cohort 3 | 200 mg Quinidine BID (Days 19 to 24): Cohort 3 | 10 mg Rosuvastatin + 0.25 mg Digoxin: Cohort 4 | 400 mg Imlunestrant + 10 mg Rosuvastatin + 0.25 mg Digoxin: Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/32 | 0/32 | 0/31 | 0/31 | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/32 | 0/32 | 0/31 | 0/31 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 2/27 | 0/27 | 3/27 | 3/27 | 9/32 | 3/32 | 0/31 | 4/31 | 0/27 | 1/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg Repaglinide: Cohort 1 (N=27) | 800 mg Imlunestrant + 0.5 mg Repaglinide: Cohort 1 (N=27) | 20 mg Omeprazole + 30 mg Dextromethorphan: Cohort 2 (N=27) | 800 mg Imlunestrant + 20 mg Omeprazole + 30 mg Dextromethorphan: Cohort 2 (N=27) | 400 mg Imlunestrant (Day 1): Cohort 3 (N=32) | 200 mg Quinidine BID (Days 15 to 17): Cohort 3 (N=32) | 400 mg Imlunestrant + 200 mg Quinidine BID (Day 18): Cohort 3 (N=31) | 200 mg Quinidine BID (Days 19 to 24): Cohort 3 (N=31) | 10 mg Rosuvastatin + 0.25 mg Digoxin: Cohort 4 (N=27) | 400 mg Imlunestrant + 10 mg Rosuvastatin + 0.25 mg Digoxin: Cohort 4 (N=26)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-06-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT05444556/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT05444556/SAP_001.pdf